CLINICAL TRIAL: NCT05808452
Title: AMO CROC Study: Self-medication and Dental Pain of Pulpal and Peri-apical Origin. Qualitative Study
Acronym: AMO-CROC
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2022 COUSSON (AMO-CROC); 2022-A01734-39 (Other: 2022-A01734-39)
Record Dates: First submitted 2023-01-18; First posted 2023-04-11 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-01

CONDITIONS: Self Medication
Keywords: Dental anxiety; Qualitative; Behaviors; Self Medication
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adult patients with dental anxiety or phobia constitute a population for which access to dental care is difficult and this situation is often associated with am low socio-economic status. According to the literature, these patients avoid conventional care, make greater use of emergency services, and self-medicate when experiencing dental pain. Moreover, little is known in the literature about the use of self medication in France, although it is known that in the general population does self medicate a lot. The objective of this study is to better understand the self-medication behaviors of patients in order to improve their care. This work aim at characterizing a population of adults in need of treatment for dental pain of pulpal or periapical origin and anxious or phobic adults in need of for dental treatment under general anesthesia. Self-medication behaviors will be studied in qualitative research during recorded interviews.

ELIGIBILITY:
Inclusion Criteria:

* Adults visiting the odontology unit for dental pain due to acute pulpitis or in need of dental treatment under general anesthesia
* Speaking French
* Able to give his/her informed consent
* Affiliated to the health social security system

Exclusion Criteria:

* Adults under guardianship or curatorship
* Adults refusing to participate

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population included in the study will be comprised of Adults visiting the odontology unit for dental pain due to acute pulpitis Adults in need of dental treatment under general anesthesia recruitment will be done during dental consultations. Their non opposotion to participate to the study will be
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
self medication behaviors description | 1 year
  Describe and understand self medication behaviors in adults visiting the odontology unit for dental pain of acute pulpal origin and in need of dental treatment under general anesthesia, via a qualitative study. A semi-structured interview will be conducted. Participants will be interviewed alone. The interviews will be conducted in face-to-face in French, following this interview guide. The data will be analyzed continuously to stop the inclusion of patients when data's saturation is reached, when no new ideas are raised. Questions about self medication related to dentistry and anxiety of the dental environment will be asked.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Yves COUSSON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (2):
- France (2):
  - CHU clermont-ferrand, Clermont-Ferrand
  - CH de Riom, Riom